CLINICAL TRIAL: NCT01887704
Title: Effect of Rotational Atherectomy on Balloon-resistant Calcified Coronary Lesion the During a Long-term Follow-up Study
Brief Title: Effect of Rotablator on Balloon Resistant Calcified Coronary Lesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, Proffesor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERBRCAL
Record Dates: First submitted 2013-06-19; First posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atherectomy, Coronary; Angioplasty, Balloon, Coronary; Stents; Aspirin; Tablets; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rotablator (Experimental): Rotablator plus conventional angioplasty and/or stenting was performed in 120 patients in the R group.
  Rotablator using 140, -160, 000 rpm, small rota burr (burr-to-artery ratio, 0.6:1), avoid drop of >5000 rpm for 5s.
  Conventional intervention will be performed in the rotablator group. All subjects were given 100 mg/day aspirin and clopidogrel (300 mg loading dose and 75 mg/day maintenance dosage) at least 24 h before the procedure. A cutting balloon, buddy wire balloon, buddy wire, or DES (including sirolimus-eluting stent, paclitaxel-eluting stent, everolimus-eluting stent,zotarolimus-eluting stent) was implemented at the discretion of the operator in both groups.
  Interventions: Device: Rotablator; Procedure: conventional angioplasty; Procedure: stenting; Device: Cutting balloon; Drug: Aspirin; Drug: Clopidogrel; Device: Paclitaxel-eluting stent; Device: zotarolimus-eluting stent; Device: Everolimus-eluting stent; Device: Sirolimus-eluting stent
- Conventional (Active Comparator): Conventional angioplasty and/or stenting was performed in 120 patients in the C group.
  Conventional intervention without rotablator was performed in the C group. All subjects were given 100 mg/day aspirin and clopidogrel (300 mg loading dose and 75 mg/day maintenance dosage) at least 24 h before the procedure. A cutting balloon, buddy wire balloon, buddy wire, or DES (including sirolimus-eluting stent, paclitaxel-eluting stent, everolimus-eluting stent,zotarolimus-eluting stent) was implemented at the discretion of the operator in both groups.
  Interventions: Procedure: conventional angioplasty; Procedure: stenting; Device: Cutting balloon; Drug: Aspirin; Drug: Clopidogrel; Device: Paclitaxel-eluting stent; Device: zotarolimus-eluting stent; Device: Everolimus-eluting stent; Device: Sirolimus-eluting stent

INTERVENTIONS:
Device: Rotablator — Rotablator, Boston Scientific, Maple Grove, MN, USA. Rotablator will be used in the Rotablator arm.
  Other Names: Rotational atherectomy; High-speed rotational atherectomy
  Arms: Rotablator
Procedure: conventional angioplasty — Conventional angioplasty was used in both arms.
  Other Names: percutaneous transluminal coronary angioplasty
Procedure: stenting — Stenting was implanted in both arms.
  Other Names: Implantation of coronary stent
Device: Cutting balloon — Flextome cutting balloon(Boston Scientific, Natick, MA, USA) was used in both arms.
  Other Names: Flextome Cutting balloon
Drug: Aspirin — Aspirin will be administrated in participants in both arms.
  Other Names: Bayaspirin, 100mg, tablet, oral, Germany
Drug: Clopidogrel — Clopidogrel will be administrated to participants in both arms.
  Other Names: Plavix, Clopidogrel Bisulfate, 100mg, tablet, oral
Device: Paclitaxel-eluting stent — Paclitaxel-eluting stent will be used in both arms.
  Other Names: Taxus
Device: zotarolimus-eluting stent — Zotarolimus-eluting stent will be implanted in participants in both arms.
  Other Names: Resolute, Medtronic CardioVascular
Device: Everolimus-eluting stent — Everolimus-eluting stent will be used in both arms.
  Other Names: Xience V
Device: Sirolimus-eluting stent — Sirolimus-eluting stent will be used in both arms.
  Other Names: Firebird, Shanghai, China

SUMMARY:
The optimal treatment of calcified coronary lesion remained to be elucidated. A Prospective, randomized controlled trial was perform to explore the immediate effect and long-term outcome of rotational atherectomy in patients with balloon resistant coronary lesion.

DETAILED DESCRIPTION:
The inclusion criteria included patients presenting drug-resistant angina pectoris who underwent balloon resistant angioplasty.

The exclusion criteria included:

1. Acute myocardial infarction within the 28 days;
2. Intolerance to aspirin, clopidogrel, contrast media, or statins;
3. Angiographic visible thrombus, or dissection;
4. Left ventricular ejection fraction (LVEF)<35%;
5. Any type of cancer
6. Hemorrhagic stroke

ELIGIBILITY:
Inclusion Criteria:

* Drug-resistant angina pectoris
* Balloon resistant and angiographic calcified coronary lesion

Exclusion Criteria:

* Acute myocardial infarction within 28 days;
* Intolerance to aspirin, clopidogrel, contrast media, or statins;
* Angiographic visible thrombus, dissection;
* LVEF <35%;
* Any type of cancer;
* Hemorrhagic stroke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events including death, myocardial infarction (MI), target vessel revascularization (TVR) and coronary artery bypass grafting | Participants will be followed for 2 years after the procedure, an expected average of 24 months.
  Follow-up study was performed by experienced doctors through telephone interviews or clinic visits at 1, 3, 6, and 12 months after the procedure, and at every 6 months thereafter. The average duration of follow up was anticipated to be 24 months.

SECONDARY OUTCOMES:
In hospital endpoints including death, periprocedural MI | In hospital endpoints were doucmented for the duration of hospital stay, an expected average 2 weeks.
  Baseline characteristics were measured on the day of admission to the hospital(baseline).An electrocardiogram was performed 2 h after the procedure. electrocardiograms were required to document any suspicious cardiac ischemic episodes. If any cardiac biomarker elevation was noted after the procedure, further measurements were performed as needed. During their hospital stays, patients were clinically monitored for the occurrence of any adverse events and the need for any additional coronary interventional treatment (In hospital endpoints including death, periprocedural MI).

OTHER OUTCOMES:
Procedural complications | Participants will be followed during the process of the procedure, an expected average of 4 hours.
  Procedural complications including death, vessel perforation, dissection, ventricular fibrillation, no reflow, side branch loss. The specific unit of measure will be number of participants with any above mentioned procedural complications.

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, MD., Study Chair
Locations (1):
- Xinguo Wang, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Chiang MH, Lee WL, Tsao CR, Chang WC, Su CS, Liu TJ, Liang KW, Ting CT. The use and clinical outcomes of rotablation in challenging cases in the drug-eluting stent era. J Chin Med Assoc. 2013 Feb;76(2):71-7. doi: 10.1016/j.jcma.2012.10.004. Epub 2012 Dec 29. PMID 23351416
- [Background] Roy P, Steinberg DH, Sushinsky SJ, Okabe T, Pinto Slottow TL, Kaneshige K, Xue Z, Satler LF, Kent KM, Suddath WO, Pichard AD, Weissman NJ, Lindsay J, Waksman R. The potential clinical utility of intravascular ultrasound guidance in patients undergoing percutaneous coronary intervention with drug-eluting stents. Eur Heart J. 2008 Aug;29(15):1851-7. doi: 10.1093/eurheartj/ehn249. Epub 2008 Jun 11. PMID 18550555